CLINICAL TRIAL: NCT00707356
Title: Vascular-Targeted Photodynamic Therapy Using WST 11 in Patients With Localized Prostate Cancer
Brief Title: Study of WST11 in Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steba Biotech S.A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN801 PCM201
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer
Keywords: Prostatic disease; genital neoplasm, male; Urogenital neoplasm; Genital disease; male; Male urogenital disease; Neoplasms; Neoplasm by site; prostatic neoplasm; Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases; Genital Neoplasms, Male; Urogenital Neoplasms; Genital Diseases; Male Urogenital Diseases; Neoplasms; Neoplasms by Site; Carcinoma | interventions — padeliporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WST11(TOOKAD® Soluble) (Experimental): Treatment with WST11-mediated VTP
  Interventions: Drug: WST11

INTERVENTIONS:
Drug: WST11 — WST11-mediated VTP will consist of the combination of a single IV administration of WST11 at doses of 2 mg/Kg,4 mg/Kg or 6 mg/kg, using 753 nm laser light at a fixed power (150mW/cm) and energy (200 J/cm) delivered through transperineal interstitial optical fibers. If deemed necessary and in consideration of the results of the patients treated with 200 J/cm, alternate power (200mW/cm) and alternate energy (300 J/cm) might be applied.The fibers are introduced into transparent needles that are positioned in the prostate under ultra sound image guidance. The number of fibers and the total light energy will be adapted to each patient, taking into account the tumor localization and the volume of the prostate.
  Other Names: WST11-mediated VTP

SUMMARY:
The aim of this clinical study is to determine the optimal treatment conditions to achieve prostate cancer tumor ablation and to assess the effects of WST11 mediated VTP treatment in patients with localized prostate cancer.

The secondary objectives is to evaluate safety and quality of life ; to assess the pharmacokinetic parameters and to model the relationship between concentration and effects; and to assess the effects, the safety and quality of life of a second WST11 VTP treatment in patients with persistent or recurrent localized prostate cancer after a first VTP;

DETAILED DESCRIPTION:
This trial is designed as a multicentre, phase II, open-labeled, single intra-venous (IV) dose study. The patient is to receive general anesthesia. WST11-mediated VTP will consist of the combination of a single IV administration of WST11 at doses of 2 mg/Kg,4mg/Kg or 6 mg/kg, using 753 nm laser light at a fixed power (150mW/cm) and energy (200 J/cm) delivered through transperineal interstitial optical fibers. If deemed necessary and in consideration of the results of the patients treated with 200 J/cm, alternate power (200mW/cm) and alternate energy (300 J/cm) might be applied after Sponsor, Steering Committee and DSMB approval.The fibers are introduced into transparent needles that are positioned in the prostate under ultra sound image guidance (using a brachytherapy like template). The tumor location is established using transrectal biopsy and MR imaging. The number of fibers and the total light energy will be adapted to each patient, taking into account the tumor localization and the volume of the prostate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer and eligible for active surveillance;
* No prior treatment for prostate cancer;
* Prostate Cancer Stage up to cT2b - N0/Nx - M0/Mx (rT2c and pT2c are acceptable);
* Gleason score ≤ 3+3 For patients characterized with prostate mapping (transperineal template guided biopsy at 5mm intervals) a secondary pattern 4 is acceptable provided that it is not present in more than 3 cores from each side of the prostate and is no more than 3 mm cancer core length.
* PSA < 10 ng/mL;

Exclusion Criteria:

* Any condition or history of illness or surgery that, in the opinion of the investigator and/or the Sponsor, might confound the results of the study or pose additional risks to the patient.
* Patients with a prior history of viral or alcoholic hepatitis, and other patients felt to be at risk for hepatotoxicity including concomitant use of potentially hepatotoxic medications or dietary supplements;
* History of non compliance with medical therapy and medical recommendations or an unwillingness or inability to complete patient self-administered questionnaires;
* Participation in a clinical study or receipt of an investigational treatment within the past 3 months;
* A history of porphyria;
* Patient with contra-indication to MRI (such as pace maker, metal prosthesis, etc.);
* All patients whose current pre-operative cardiac evaluation does not show their fitness for a procedure requiring general anesthesia;
* Patients with a history of inflammatory bowel disease or other factors which may increase the risk of fistula formation;
* Men who have received any hormonal manipulation (excluding 5-alpha reductase inhibitors) or androgen supplements within the previous 6 months;
* Men previously treated by radiation therapy (external therapy or brachytherapy) or chemotherapy or any therapy for prostate cancer;
* Men who have received or are receiving chemotherapy for prostate carcinoma or other significant cancer;
* Men who have undergone previous TURP (trans-urethral resection of the prostate);
* Men who are currently receiving any medications having potential photosensitizing effects (e.g. tetracyclines, sulfonamides, phenothiazines, sulfonylurea hypoglycemic agents, thiazide diuretics and griseofulvin);
* Men who are receiving anticoagulant drugs (e.g.: coumadin, warfarin)
* Patient who stopped long term treatment of acetylsalicylic acid (aspirin) or other anti platelets agents less than 15 days before the procedure;
* Patient suspected of Disseminated Intravascular Coagulation (DIC) as defined by the presence of three out of the five following criteria: platelets <LLN, PT >ULN,aPTT >ULN, fibrinogen<LLN, D-Dimer >ULN;
* A history of sun hypersensitivity or photosensitive dermatitis;
* Renal disorders (blood creatinine > 1.5 x ULN) or known post mictional residue > 150cc;
* Hepatic disorders (transaminases > ULN, bilirubin > ULN). In case of slight abnormalities, another exam should be performed. If the results are within normal ranges, then the patient can be included;
* Hematological disorders (white cells < 2500/mm3, neutrophils < 1500/mm3, platelets < 140.000/mm3, Hb < 8 g/dl);

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Negative biopsy in the treated lobe | Month 6

SECONDARY OUTCOMES:
Volume of the hypoperfusion area shown by dynamic gadolinium MRI . Serum PSA levels and PSA changes . Adverse Events, ECG (12-lead), vital signs, clinical laboratory evaluations, physical examination Quality of Life:•IPSS •IIEF | Day 7; Month 1 ;3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Mark EMBERTON, Professor, Principal Investigator — Urology Directorate
Locations (8):
- University Health Network-Princess Margaret Hospital, Toronto, Canada
- France (4):
  - Centre Hospitalier Universitaire, Angers
  - Hôpital Bocage-CHU, Dijon
  - Hôpital Claude Huriez, Lille
  - Institut Mutualiste Montsouris(IMM), Paris
- United Kingdom (3):
  - Frimley Park Hospital NHS Trust, Frimley
  - Kings College Hospital(KCH), London
  - Urology Directorate, London

IPD SHARING:
Plan to Share IPD: Yes
The data are available in case report form for each patient

REFERENCES:
- [Result] Moore CM, Azzouzi AR, Barret E, Villers A, Muir GH, Barber NJ, Bott S, Trachtenberg J, Arumainayagam N, Gaillac B, Allen C, Schertz A, Emberton M. Determination of optimal drug dose and light dose index to achieve minimally invasive focal ablation of localised prostate cancer using WST11-vascular-targeted photodynamic (VTP) therapy. BJU Int. 2015 Dec;116(6):888-96. doi: 10.1111/bju.12816. Epub 2015 Apr 21. PMID 24841929
- [Derived] Azzouzi AR, Lebdai S, Benzaghou F, Stief C. Vascular-targeted photodynamic therapy with TOOKAD(R) Soluble in localized prostate cancer: standardization of the procedure. World J Urol. 2015 Jul;33(7):937-44. doi: 10.1007/s00345-015-1535-2. Epub 2015 Mar 19. PMID 25786708
- [Derived] Azzouzi AR, Barret E, Bennet J, Moore C, Taneja S, Muir G, Villers A, Coleman J, Allen C, Scherz A, Emberton M. TOOKAD(R) Soluble focal therapy: pooled analysis of three phase II studies assessing the minimally invasive ablation of localized prostate cancer. World J Urol. 2015 Jul;33(7):945-53. doi: 10.1007/s00345-015-1505-8. Epub 2015 Feb 25. PMID 25712310
- [Derived] Lebdai S, Villers A, Barret E, Nedelcu C, Bigot P, Azzouzi AR. Feasibility, safety, and efficacy of salvage radical prostatectomy after Tookad(R) Soluble focal treatment for localized prostate cancer. World J Urol. 2015 Jul;33(7):965-71. doi: 10.1007/s00345-015-1493-8. Epub 2015 Jan 23. PMID 25614256
- [Derived] Colin P, Estevez JP, Betrouni N, Ouzzane A, Puech P, Leroy X, Biserte J, Villers A, Mordon S. [Photodynamic therapy and prostate cancer]. Prog Urol. 2011 Feb;21(2):85-92. doi: 10.1016/j.purol.2010.07.018. Epub 2010 Sep 17. French. PMID 21296274